CLINICAL TRIAL: NCT06641999
Title: A Prospective, Multicentric, Feasibility Investigation to Assess the Effect of the Tinnitus Implant on Tinnitus Loudness in Adults With Moderate to Severe Chronic Tinnitus Accompanied by Normal Hearing to Moderately Severe Hearing Loss.
Brief Title: Evaluating How a Tinnitus Implant Affects Tinnitus Loudness in Adults With Chronic Tinnitus and Varying Levels of Hearing Loss
Acronym: TINIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI5856
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Tinnitus; Hearing Loss, Bilateral or Unilateral; Normal Hearing
Keywords: tinnitus; cochlear implant
MeSH Terms: conditions — Tinnitus; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tinnitus Implant System (Experimental): Tinnitus Implant
  Interventions: Device: Tinnitus Implant System

INTERVENTIONS:
Device: Tinnitus Implant System — Implanted with Tinnitus Implant System: Active Implantable Medical Device

SUMMARY:
This study will test an experimental Tinnitus Implant System that consists of a cochlear implant, sound processor and programming software. The Tinnitus implant is surgically placed under the skin just behind the ear in the mastoid bone. It has an electrode that extends from the implant into the promontory bone of the cochlea which emits electrical signals that stimulate the auditory nerve. The sound processor is worn behind the ear and powers the implant via the coil. The study will be conducted in adults with moderate to severe chronic tinnitus who have normal hearing to moderately severe hearing loss in the inner ear. The study participants will undergo a series of tests that include evaluations of tinnitus loudness and annoyance, and self-reported questionnaires on their tinnitus and general health.

ELIGIBILITY:
Inclusion criteria

* 18 years or older.
* Normal hearing to moderately severe sensorineural hearing loss defined as a pure tone average (PTA) at 500, 1000, 2000 and 4000 Hz less than 65 dB HL in both ears (separately) and best-aided phoneme recognition score more than or equal to 80% in both ears (separately).
* Unilateral or asymmetric subjective (no pulsatile) tinnitus. In case of asymmetric tinnitus, the worst ear must be implanted.
* Tinnitus duration of at least 6 months.
* Severe tinnitus loudness determined by a. VAS-L score in the severe range i.e. 50-100/100 b. TFI score in the severe range i.e. 52-90/100
* Tinnitus that is intractable and has not been ameliorated satisfactorily by standard of care such as CBT or hearing aid, when such interventions are potentially clinically indicated.
* Clinically significant reduction in VAS-L score (≥ 15/100 points) in response to trans-tympanic promontory stimulation
* Willing and able to provide written informed consent.
* Medically able to use the device and to undergo general anaesthesia for implantation taking into account their medical condition, contraindications and surgical risks.
* Dutch language proficiency

Exclusion Criteria:

* Pulsatile tinnitus.
* Any anatomical or structural abnormalities of the inner ear, cochlear nerve, or brainstem that would negatively impact response to study intervention (determined in a temporal bone CT and if necessary (e.g. possibility of vestibular/acoustic schwannoma) by a MRI scan of the head (of sufficient quality at the discretion of the investigator) not more than five years old at the time of enrolment
* Medical contraindications limiting correct placement, activation, or treatment (determined by medical history; contraindications include brain or major ear surgery, brain or temporal bone tumor(s), recurrent ear infections within the last year, otosclerosis, prior major head trauma that results in sudden injury that causes damage to the brain and results in lasting cognitive impairment).
* Any medical condition, including mental illness or substance abuse, deemed by the Investigator to likely interfere with a patient's ability to sign informed consent, cooperate and/or participate in the study, or interfere with the interpretation of the results (incl. pregnant or breastfeeding women or patients with unrealistic expectations).
* Presence of clinically diagnosed depression or anxiety determined by a psychological state evaluation (if PHQ-9 > 9 or GAD-7 > 9).
* Active (currently or within two months prior to enrolment) use of medications (taking regularly scheduled antidepressant, anxiolytic, antipsychotic or antiepileptic medications, or other neuromodulator agents) or other tinnitus treatments.
* It is permissible to include people who use such medications at lower doses as a sleep aid or for people who intermittently use such medications for situational anxiety (e.g., Ativan before airplane travel). A change in medication during the trial should be avoided.
* It is permissible to include people who prefer to use a hearing aid to amplify ipsilateral hearing loss. The start of using a hearing aid during the trial should be avoided.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 60 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in tinnitus loudness from baseline to 6 months post-activation of the Tinnitus Implant System | Pre-operative baseline to 6 months post Tinnitus Implant System activation
  Self-reported tinnitus loudness as measured on the Visual Analogue Scale-Loudness (VAS-L) where 0 is equivalent to absence of tinnitus and 100 indicates tinnitus of the greatest loudness severity

SECONDARY OUTCOMES:
Reported device or procedure related adverse events and harms | Pre-operative baseline to 6 months post Tinnitus Implant System activation
  Number of device and procedure-related adverse events and reported harms
Mean change in tinnitus annoyance from baseline to 6 months post activation of the Tinnitus Implant System | Pre-operative baseline to 6 months post Tinnitus Implant System activation
  Self-reported tinnitus loudness as measured on the Visual Analogue Scale-Annoyance (VAS-A) where 0 is equivalent to absence of tinnitus and 100 indicates tinnitus of the greatest annoyance severity
Mean change in tinnitus perception from baseline to 6 months post activation of the Tinnitus Implant System | Pre-operative baseline to 6 months post Tinnitus Implant System activation
  Self-reporting on the Tinnitus Functional Index (TFI) questionnaire
Change in self-reported matches of tinnitus pitch and loudness to acoustic stimuli | Pre-operative baseline, activation (Implant activation is approximately 10 weeks after surgical implantation of Tinnitus implant), 3 months post activation, 6 months post activation
  Patient reported matching of tinnitus pitch (Hz) and loudness (dB SPL) with acoustic stimuli
Mean change in health-related quality of life with Tinnitus Implant System | 6 months post Tinnitus Implant System activation
  Score of Glasgow Benefit Inventory (GBI) questionnaire
Mean change in health status with Tinnitus Implant System | At 6 months post Tinnitus Implant System activation
  Score of Patient Global Impression of Change (PGIC) questionnaire
Mean change in speech perception in quiet from baseline to 6 months post-activation | Pre-operative baseline to 6 months post Tinnitus Implant System activation
  Word recognition in quiet presented at 65 dB SPL in the unaided condition
Mean change in hearing thresholds from baseline to 6 months post-activation | Pre-operative baseline to 6 months post Tinnitus Implant System activation
  Bone conduction thresholds (dB HL) at any tested frequency (0.25, 0.5, 1, 1.5, 2, 4 kHz) from baseline to 6 months post-activation in the implanted ear

CONTACTS AND LOCATIONS:
Overall Officials: Remo Arts, Study Director — Cochlear
Locations (2):
- Antwerp University Hospital (UZA), Edegem, Belgium, Belgium
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No